CLINICAL TRIAL: NCT02984891
Title: Dual Imaging Using High-definition Intravascular Ultrasound and Optical Coherence Tomography to Guide Percutaneous Coronary Intervention
Brief Title: Optical Coherence Tomography (OCT) Intravascular Ultrasound (IVUS) Dual Imaging
Status: Terminated | Type: Observational
Why Stopped: Slow enrollment
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: AAAQ8295
Record Dates: First submitted 2016-12-05; First posted 2016-12-07 (Estimated); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Coronary Artery Disease (CAD)
Keywords: Intravascular ultrasound; Optical coherence tomography
MeSH Terms: conditions — Coronary Artery Disease | interventions — Tomography, Optical Coherence; Ultrasonography, Interventional

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treatment: Intravascular Ultrasound (IVUS) and Optical Coherence Tomography (OCT) will be used in patients with coronary artery disease.
  Interventions: Procedure: Optical Coherence Tomography (OCT); Procedure: Intravascular Ultrasound (IVUS)

INTERVENTIONS:
Procedure: Optical Coherence Tomography (OCT) — Procedure will be performed using the OCT Dragonfly catheter is a hydrophilic-coated catheter that uses infrared light with a central wavelength between 1,250 and 1,350 nm. Axial resolution with OCT is 10-20 microns, and maximum tissue penetration with OCT is approximately 1.5 mm-3 mm.
  Other Names: OCT
Procedure: Intravascular Ultrasound (IVUS) — Procedure will be performed using the IVUS Kodama catheter is a hydrophilic-coated catheter that used high-fidelity ultrasound transmission to capture high-definition images of coronary artery anatomy. It uses ultrasound waves with a frequency of 40 or 60 MHz, as opposed to 20 MHz in conventional IVUS, to improve resolution while optimizing tissue penetration. It provides axial resolution of < 40 microns and tissue penetration of 10 mm.
  Other Names: IVUS

SUMMARY:
Both intravascular ultrasound (IVUS) and optical coherence tomography (OCT) are standardly used and have been extensively studied separately to guide percutaneous coronary intervention and improve long-term outcomes. In this study, the investigators aim to directly compare high-definition IVUS images to OCT in the same patients to determine the differences between each modality as they relate to imaging coronary pathology, with the goal of determining which modality is most appropriate in particular clinical scenarios.

DETAILED DESCRIPTION:
Intravascular ultrasound (IVUS) is an imaging modality that uses ultrasound waves to allow for detailed evaluation of coronary atherosclerotic plaques and the vascular response to coronary interventional devices to guide stent placement during percutaneous coronary intervention. Current conventional IVUS catheters emit ultrasound waves ranging from 20-40 megahertz (mHz), and more recently released high-definition IVUS catheters emit sound waves at 60 mHz, allowing for better image quality, quantitative accuracy, and precision in measurements.

Optical coherence tomography (OCT) is an alternative imaging modality used for similar purposes as IVUS, using a single optical fiber that emits infrared light to image the coronary artery. OCT uses light in the infrared spectrum with a central wavelength between 1,250 and 1,350 nm. Axial resolution with OCT is 10-20 microns, whereas it is typically 100-200 microns with IVUS. Thus, OCT allows for better image resolution, but this comes at the expense of tissue penetration.

ELIGIBILITY:
Inclusion criteria:

* Undergone diagnostic coronary angiography
* Evidence of coronary pathology that requires further imaging to guide treatment

Exclusion criteria:

Significant renal insufficiency

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients included in the study will be those with coronary artery disease who are scheduled to undergo standard angiography in the cardiac catheterization lab.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2016-10-06 (Actual); Primary Completion 2018-06-27 (Actual); Study Completion 2018-06-27 (Actual)

PRIMARY OUTCOMES:
Lumen area | Up to 1 hour
Luminal diameter | Up to 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Ziad A. Ali, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No